CLINICAL TRIAL: NCT06665984
Title: Greater Houston Area Pediatric Bipolar Registry
Acronym: GHAPBR
Status: Recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: John S. Dunn Foundation (Unknown)
Responsible Party: Principal Investigator, Jair Soares, Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-20-0329
Record Dates: First submitted 2023-08-04; First posted 2024-10-30 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Pediatric Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 19 Years
Biospecimen Retention: Samples With DNA — Approximately 2ml of Saliva will be collected and processed for DNA. Blood will be collected and plasma and peripheral blood mononuclear cells (PBMCs) will be isolated
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Bipolar Patients
- Offspring of Bipolar Parents
- Healthy Control Subjects

SUMMARY:
The purpose of this study is to perform a comprehensive research assessment of children and adolescents who meet The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) criteria for Bipolar Disorder (BD) , offspring of a parent with BD, and healthy controls (HC), to obtain blood samples and saliva samples from each subject to allow the evaluation for BD biomarkers and genetic information, to notify participants about future research studies they may qualify for , to recommend follow-up with an outpatient provider if needed and to use magnetic resonance imaging (MRI) (structural MRI and diffusion tensor imaging) to investigate brain structures and relevant pathways associated with mood and behavioral regulation, conversion from softer forms of the BD spectrum (BD-NOS) to harder forms (BD-I and BD-II) and possible early identification.

ELIGIBILITY:
Inclusion Criteria for bipolar patients or offspring of bipolar parents:

* Any current mood state (in the case of bipolar subjects)
* For bipolar patients: DSM-V criteria for BD type I, BD type II, or BD NOS, as per the administration of the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID)
* For the offspring of bipolar parents: at least one parent meeting DSM-V criteria for BD type I or BD type II, or BD NOS as per the administration of the MINI Adult

Exclusion Criteria for bipolar patients or offspring of bipolar parents:

* Autism Spectrum Disorder (ASD)
* Developmental Intellectual Disorder
* Severe Neurological Disorder that affects cognitive status (e.g., epilepsy, traumatic brain injury, tubular sclerosis)
* Schizophrenia
* Uncontrolled or severe medical problem per investigator judgment
* For the offspring: parents with a history of any brain diseases, including seizures, stroke, meningitis, encephalitis, dementia, and other degenerative brain diseases; parents with a history of intellectual disability

Exclusion Criteria for healthy control subjects:

* Any Psychiatric Diagnosis
* Any family history of Bipolar Disorder, Psychotic Disorder, Schizophrenia, or Schizoaffective disorder in a first-degree relative
* Any family history of a neurological condition in a first-degree relative.
* Mental Retardation/Intellectual Disability
* Severe Neurological Disorder that affects cognitive status (e.g., epilepsy, traumatic brain injury, tubular sclerosis)
* Schizophrenia
* Uncontrolled or severe medical problem per investigator judgement

Exclusion criteria for annual visits:

* Autism Spectrum Disorders (ASD)
* Intellectual Developmental Disorder
* Severe Neurological Disorder that affects cognitive status (e.g., epilepsy, traumatic brain injury, tubular sclerosis)
* Schizophrenia
* Uncontrolled or severe medical problem per investigator judgement

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects will be recruited from the Harris County Psychiatric Center, Harris Center for Mental Health, Texana Behavioral Healthcare Clinic, and UT Child and Adolescent Outpatient Psychiatry Clinic at Behavioral Science Campus, community referrals, referrals from other health providers, as well as self-referrals.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2027-12-06 (Estimated); Study Completion 2046-12-06 (Estimated)

PRIMARY OUTCOMES:
Positive Identification of Bipolar Disorder as Assessed by Mini-International Neuropsychiatric Interview for Children and Adolescents (MINI Kid 7.2) (child) | baseline, annually until participant turns 25 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Jair C Soares, M.D. PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No